CLINICAL TRIAL: NCT02452099
Title: Impact of Different DMSO Concentrations in Cryopreservation Mixture on Hematopoietic Recovery After Autologous Transplantation of Hematopoietic Stem Cells.
Brief Title: Impact of DMSO Concentrations on Hematopoietic Recovery After Autologous HSC Transplantation.
Acronym: DMSOconc3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Principal Investigator, Sebastian Giebel, Prof., MD, Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COI-DMSO-01
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Myeloma; Lymphomas; Leukemias
Keywords: DMSO; cryopreservation; autologous transplantation; hematopoietic stem cells; hematological malignancies
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Leukemia; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5% DMSO (Other)
  Interventions: Procedure: Cryopreservation of HSCs using 5% DMSO concentration
- 7.5% DMSO (Other)
  Interventions: Procedure: Cryopreservation of HSCs using 7,5% DMSO concentration
- 10% DMSO (Other)
  Interventions: Procedure: Cryopreservation of HSCs using 10% DMSO concentration

INTERVENTIONS:
Procedure: Cryopreservation of HSCs using 5% DMSO concentration — Cryopreservation of HSCs obtained by leukapheresis will be performed using 5% DMSO concentration.
  Arms: 5% DMSO
Procedure: Cryopreservation of HSCs using 7,5% DMSO concentration — Cryopreservation of HSCs obtained by leukapheresis will be performed using 7,5% DMSO concentration.
  Arms: 7.5% DMSO
Procedure: Cryopreservation of HSCs using 10% DMSO concentration — Cryopreservation of HSCs obtained by leukapheresis will be performed using 10% DMSO concentration.
  Arms: 10% DMSO

SUMMARY:
The main aim of the study was to evaluate the clinical impact of different DMSO concentrations in cryopreservation mixture (5%, 7.5%, 10%) on reconstitution of hematopoiesis after autologous hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
The procedure of autologous hematopoietic stem cell (HSC) transplantation requires cryopreservation of HSCs. Addition of DMSO (dimethyl sulfoxide) is necessary to secure the viability of such cells, but this cryoprotectant is potentially toxic to stem cell recipient. The concentrations of DMSO in cryopreservation mixture vary strongly between protocols in different transplant centers. Usually, the HSCs are stored in mixtures containing 10% DMSO, but there is no sufficient evidence that this concentration of DMSO is indeed optimal.

The main aim of the study is to evaluate the clinical impact of reduction of DMSO concentration in cryopreservation mixture on engraftment after autologous hematopoietic stem cell transplantation. 150 consecutive patients will be randomly assigned to one of three study arms (50 patients each). HSCs obtained by leukapheresis will be cryopreserved in three concentrations of DMSO: 5%, 7.5%, 10%, respectively. Evaluation of the mixtures will be carried out by monitoring reconstitution of hematopoiesis and the frequency the side effects in patients. The most important aspect of our evaluation will be the speed of neutrophil recovery after transplantation (defined by the first day, when absolute neutrophil count in peripheral blood will be higher than 0.5 G/L). The investigators will also evaluate the toxicity of cell suspension by monitoring the frequency of infusion-related adverse events (like nausea or vomiting) during infusion and 24 hours after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological malignancies or solid tumors, refered for autologous HSC transplantation
* Written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The median time to neutrophils recovery after autoHSC transplantation. | The first from 3 consecutive days, on which absolute neutrophil count in peripheral blood will be higher than 0.5 G/L

SECONDARY OUTCOMES:
The median time to platelets recovery after autoHSC transplantation. | The first from 3 consecutive days, on which platelet count in peripheral blood will be higher than 20 G/L, without platelet transfusion 7 days prior.
Adverse reactions related with transplantation procedure | 24 hours after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- MSC Memorial CAncer Center and Institute of Oncology, Gliwice, Poland

REFERENCES:
- [Result] Smagur A, Mitrus I, Ciomber A, Panczyniak K, Fidyk W, Sadus-Wojciechowska M, Holowiecki J, Giebel S. Comparison of the cryoprotective solutions based on human albumin vs. autologous plasma: its effect on cell recovery, clonogenic potential of peripheral blood hematopoietic progenitor cells and engraftment after autologous transplantation. Vox Sang. 2015 May;108(4):417-24. doi: 10.1111/vox.12238. Epub 2015 Mar 6. PMID 25753814
- [Result] Mitrus I, Smagur A, Giebel S, Gliwinska J, Prokop M, Glowala-Kosinska M, Chwieduk A, Sadus-Wojciechowska M, Tukiendorf A, Holowiecki J. A faster reconstitution of hematopoiesis after autologous transplantation of hematopoietic cells cryopreserved in 7.5% dimethyl sulfoxide if compared to 10% dimethyl sulfoxide containing medium. Cryobiology. 2013 Dec;67(3):327-31. doi: 10.1016/j.cryobiol.2013.09.167. Epub 2013 Oct 11. PMID 24125911
- [Result] Smagur A, Mitrus I, Giebel S, Sadus-Wojciechowska M, Najda J, Kruzel T, Czerw T, Gliwinska J, Prokop M, Glowala-Kosinska M, Chwieduk A, Holowiecki J. Impact of different dimethyl sulphoxide concentrations on cell recovery, viability and clonogenic potential of cryopreserved peripheral blood hematopoietic stem and progenitor cells. Vox Sang. 2013 Apr;104(3):240-7. doi: 10.1111/j.1423-0410.2012.01657.x. Epub 2012 Oct 9. PMID 23046417